CLINICAL TRIAL: NCT04976322
Title: A Multicenter, Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of Dapirolizumab Pegol Treatment in Study Participants With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety and Tolerability of Dapirolizumab Pegol in Study Participants With Systemic Lupus Erythematosus
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL0046; 2019-003409-83 (EudraCT Number); U1111-1293-7098 (Other: World Health Organization (WHO)); 2023-506368-14 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Dapirolizumab pegol; SLE; DZP
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — dapirolizumab pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapirolizumab pegol (Experimental): Subjects will receive dapriolizumab pegol throughout the Treatment Period.
  Interventions: Drug: Dapirolizumab pegol

INTERVENTIONS:
Drug: Dapirolizumab pegol — Subjects will receive dapirolizumab pegol at prespecified time-points.
  Other Names: DZP; CDP7657

SUMMARY:
The purpose of this study is to evaluate long-term safety and tolerability of dapirolizumab pegol treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant could, in the opinion of the Investigator, benefit from long-term dapirolizumab pegol (DZP) treatment
* The participant completed one of the parent studies within 4 weeks prior to entry to this study

Exclusion Criteria:

- Study participant has any medical or psychiatric condition (including conditions due to neuropsychiatric systemic lupus erythematosus (SLE)) that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study. This includes study participants with a life-threatening condition or ongoing malignancies at the start of the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2030-08-07 (Estimated); Study Completion 2030-08-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) during the study | From Baseline (Day 1) until Safety Follow-Up (up to Week 110)
  Treatment-emergent adverse events (TEAEs) are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment.
Incidence of serious treatment-emergent adverse events during the study | From Baseline (Day 1) until Safety Follow-Up (up to Week 110)
  A serious treatment-emergent adverse event (serious TEAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent disability/incapacity
  * Is a congenital anomaly or birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of treatment-emergent adverse events (TEAEs) leading to permanent dapirolizumab pegol discontinuation | From Baseline (Day 1) until Safety Follow-Up (up to Week 110)
  Treatment-emergent adverse events (TEAEs) are any untoward medical incidence in a subject during administered study treatment, and leading to permanent drug discontinuation whether or not these events are related to study treatment.

SECONDARY OUTCOMES:
Achievement of prevention of severe BILAG flares (severe BILAG flare-free) through Week 24 | Week 24
  BILAG severe flare is defined as a new British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) Grade A since previous visit in any system due to individual items that are new or worse qualifying for the Grade A (Isenberg et al, 2011). Determination of items that are new or worse qualifying for the Grade A will be according to the supplementary information for the numerical scoring of the BILAG-2004 index (Yee et al, 2010).
Achievement of prevention of severe BILAG flares (severe BILAG flare-free) through Week 52 | Week 52
  BILAG severe flare is defined as a new British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) Grade A since previous visit in any system due to individual items that are new or worse qualifying for the Grade A (Isenberg et al, 2011). Determination of items that are new or worse qualifying for the Grade A will be according to the supplementary information for the numerical scoring of the BILAG-2004 index (Yee et al, 2010).
Achievement of prevention of severe BILAG flares (severe BILAG flare-free) through Week 104 | Week 104
  BILAG severe flare is defined as a new British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) Grade A since previous visit in any system due to individual items that are new or worse qualifying for the Grade A (Isenberg et al, 2011). Determination of items that are new or worse qualifying for the Grade A will be according to the supplementary information for the numerical scoring of the BILAG-2004 index (Yee et al, 2010).
Achievement of LLDAS at ≥50% of all visits | From Baseline (Day 1) until End of Treatment (Week 104)
  Low lupus disease activity state (LLDAS) is defined as:
  * No significant disease activity as per SLEDAI-2K and BILAG 2004 (SLEDAI-2K score ≤4 with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever)
  * No new and/or worsening disease activity defined as no SLEDAI-2K component documented as present that was not documented present at previous visit
  * PGA ≤33 mm
  * Prednisone equivalent systemic dose for systemic lupus erythematosus (SLE) indication ≤7.5 mg per day
  * Stable standard maintenance doses of immunosuppressive drugs as allowed by protocol
Achievement of BICLA response at Week 24 | Week 24
  A study participant is considered to be a BILAG 2004-based Composite Lupus Assessment (BICLA) responder if all of the following is fulfilled:
  1. British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤1 new B.); and
  2. No worsening in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score compared to Baseline Visit (defined as no increase in SLEDAI-2K total score); and
  3. No worsening in the Physician's Global Assessment of Disease (PGA) compared to Baseline Visit defined as ≤10 mm increase on a 100 mm visual analog scale
  The parent studies Baseline will be used as reference point.
Achievement of BICLA response at Week 52 | Week 52
  A study participant is considered to be a BICLA responder if all of the following is fulfilled:
  1. BILAG 2004 improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤1 new B.); and
  2. No worsening in the SLEDAI-2K total score compared to Baseline Visit (defined as no increase in SLEDAI-2K total score); and
  3. No worsening in the PGA compared to Baseline Visit defined as ≤10 mm increase on a 100 mm visual analog scale
  The parent studies Baseline will be used as reference point.
Achievement of BICLA response at Week 104 | Week 104
  A study participant is considered to be a BICLA responder if all of the following is fulfilled:
  1. BILAG 2004 improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤1 new B.); and
  2. No worsening in the SLEDAI-2K total score compared to Baseline Visit (defined as no increase in SLEDAI-2K total score); and
  3. No worsening in the PGA compared to Baseline Visit defined as ≤10 mm increase on a 100 mm visual analog scale
  The parent studies Baseline will be used as reference point.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (98):
- United States (26):
  - Sl0046 50140, Birmingham, Alabama
  - Sl0046 50328, Tucson, Arizona
  - Sl0046 50383, Beverly Hills, California
  - Sl0046 50275, La Palma, California
  - Sl0046 50316, San Leandro, California
  - Sl0046 50339, Denver, Colorado
  - Sl0046 50239, Brandon, Florida
  - Sl0046 50362, Gainesville, Florida
  - Sl0046 50681, Miami, Florida
  - Sl0046 50059, Ormond Beach, Florida
  - Sl0046 50324, Plantation, Florida
  - Sl0046 50329, Tampa, Florida
  - Sl0046 50368, Atlanta, Georgia
  - Sl0046 50240, Idaho Falls, Idaho
  - Sl0046 50474, Hopkinsville, Kentucky
  - Sl0046 50285, Lake Charles, Louisiana
  - Sl0046 50015, Hagerstown, Maryland
  - Sl0046 50219, Detroit, Michigan
  - Sl0046 50273, Las Vegas, Nevada
  - Sl0046 50366, Canton, New York
  - Sl0046 50334, New York, New York
  - Sl0046 50238, Charlotte, North Carolina
  - Sl0046 50147, Hershey, Pennsylvania
  - Sl0046 50001, Jackson, Tennessee
  - Sl0046 50418, Colleyville, Texas
  - Sl0046 50050, Beckley, West Virginia
- Argentina (6):
  - Sl0046 60002, Buenos Aires
  - Sl0046 60029, Mendoza
  - Sl0046 60003, Quilmes
  - Sl0046 60022, Quilmes
  - Sl0046 60011, San Juan
  - Sl0046 60014, San Miguel de Tucumán
- Sl0046 40123, Brussels, Belgium
- Bulgaria (2):
  - Sl0046 40189, Plovdiv
  - Sl0046 40380, Sofia
- Canada (4):
  - Sl0046 50374, Calgary
  - Sl0046 50337, Edmonton AB
  - Sl0046 50259, Rimouski
  - Sl0046 50045, Toronto
- Chile (2):
  - Sl0046 60015, Santiago
  - Sl0046 60018, Santiago
- Colombia (7):
  - Sl0046 60013, Barranquilla
  - Sl0046 60019, Barranquilla
  - Sl0046 60006, Bogotá
  - Sl0046 60027, Bogotá
  - Sl0046 60016, Bucaramanga
  - Sl0046 60007, Chía
  - Sl0046 60031, Montería
- Sl0046 40066, Prague, Czechia
- Germany (5):
  - Sl0046 40386, Cologne
  - Sl0046 40072, Freiburg im Breisgau
  - Sl0046 40027, Herne
  - Sl0046 40078, Leipzig
  - Sl0046 40402, Tübingen
- Greece (4):
  - Sl0046 40378, Athens
  - Sl0046 40501, Athens
  - Sl0046 40377, Crete
  - Sl0046 40507, Larissa
- Hungary (4):
  - Sl0046 40412, Budapest
  - Sl0046 40411, Debrecen
  - Sl0046 40031, Szeged
  - Sl0046 40499, Székesfehérvár
- Italy (2):
  - Sl0046 40084, Catania
  - Sl0046 40448, Milan
- Mexico (6):
  - Sl0046 50317, Chihuahua City
  - Sl0046 50250, Cuernavaca
  - Sl0046 50249, Guadalajara
  - Sl0046 50271, León
  - Sl0046 50252, Mérida
  - Sl0046 50251, Monterrey
- Peru (2):
  - Sl0046 60009, Lima
  - Sl0046 60023, Lima
- Philippines (2):
  - Sl0046 20182, Davao City
  - Sl0046 20181, Makati
- Poland (11):
  - Sl0046 40482, Bialystok
  - Sl0046 40119, Bydgoszcz
  - Sl0046 40398, Katowice
  - Sl0046 40502, Krakow
  - Sl0046 40151, Lublin
  - Sl0046 40044, Poznan
  - Sl0046 40090, Poznan
  - Sl0046 40097, Warsaw
  - Sl0046 40098, Warsaw
  - Sl0046 40397, Wroclaw
  - Sl0046 40481, Wroclaw
- Sl0046 40382, Galati, Romania
- Serbia (2):
  - Sl0046 40393, Belgrade
  - Sl0046 40461, Belgrade
- South Korea (2):
  - Sl0046 20108, Incheon
  - Sl0046 20104, Seoul
- Spain (4):
  - Sl0046 40160, Barcelona
  - Sl0046 40341, Málaga
  - Sl0046 40101, Sabadell
  - Sl0046 40099, Vigo
- Taiwan (4):
  - Sl0046 20113, Taichung
  - Sl0046 20142, Taichung
  - Sl0046 20095, Taipei
  - Sl0046 20082, Taiyuan

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org